CLINICAL TRIAL: NCT02503150
Title: Phase III Trial of Antigen Pulsed Dendritic Cells (APDC) Combined With Chemotherapy in Metastatic Colorectal Cancer
Brief Title: Trial of Antigen Pulsed Dendritic Cells (APDC) in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Military Medical University (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Changhai Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Fudan University (Other); Shanghai Changzheng Hospital (Other); Zhejiang Cancer Hospital (Other); Chinese PLA General Hospital (Other); Peking University Cancer Hospital & Institute (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); RenJi Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First People's Hospital of Hangzhou (Other); 307 Hospital of PLA (Other); Huashan Hospital (Other); Ruijin Hospital (Other); Shanghai Haixin Biotechnology Co. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMMU, Shanghai
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Tumor Therapeutic Vaccine; Dendritic Cell
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APDC + Chemotherapy (Experimental): Patients in Arm APDC + Chemotherapy will receive APDC combined with chemotherapy.
  Interventions: Biological: APDC + Chemotherapy
- Chemotherapy (Active Comparator): Patients in Arm Chemotherapy will receive chemotherapy only.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Biological: APDC + Chemotherapy — Patients in Arm APDC+Chemotherapy receive maximum 12 cycles (14days/cycle) mFOLFOX6 chemotherapy. Each cycle chemotherapy consist of Oxaliplatin at 85mg/ m2 infused for 2 hours only on day 1,and Leucovorin at 400 mg/m2 was administered intravenously for 2 hours, followed by continuous intravenous administration of 5-Fluorouracil at 400 mg/m2 (2.4g/m2 for 46 hours).On day 8 of cycle1-3 and 7-9, patients also receive APDC vaccine infusion in 100ml saline. After 12 cycles, patients in Arm APDC+chemotherapy will receive 5-Fluorouracil /Leucovorin (Leucovorin at 400 mg/m2/day administered intravenously for 2 hours, intravenous bolus of 5-Fluorouracil at 400 mg/m2 , followed by continuous intravenous administration of 5-Fluorouracil at 1200 mg/m2/d for 2 days, repeated every 2 weeks) plus APDC therapy (once every 3 months). Treatments will continue unless disease progression, intolerable toxicity or patients withdrawal).
  Arms: APDC + Chemotherapy
Drug: Chemotherapy — Patients in Arm Chemotherapy receive maximum 12cycles (14days/cycle) mFOLFOX6 chemotherapy. Each cycle chemotherapy consist of Oxaliplatin at 85mg/ m2 infused for 2 hours only on day 1, and Leucovorin at 400 mg/m2 was administered intravenously for 2 hours, followed by continuous intravenous administration of 5-Fluorouracil at 400 mg/m2 (2.4g/m2 for 46 hours). After 12 cycles, patients in Arm chemotherapy will receive only 5-Fluorouracil /Leucovorin (Leucovorin at 400 mg/m2/day administered intravenously for 2 hours, intravenous bolus of 5-Fluorouracil at 400 mg/m2 , followed by continuous intravenous administration of 5-Fluorouracil at 1200 mg/m2/d for 2 days, repeated every 2 weeks). Treatments will continue unless disease progression, intolerable toxicity or patients withdrawal).
  Arms: Chemotherapy

SUMMARY:
This trial is to compare the efficacy and safety of modified FOLFOX6 [mFOLFOX6, a specific chemotherapy regimen of Oxaliplatin ,5-Fluorouracil and Leucovorin] chemotherapy plus Antigen Pulsed Dendritic Cells (APDC，a kind of autologous tumor lysates pulsed human dendritic cells vaccine) with modified chemotherapy alone in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Metastatic colorectal cancer (CRC) patients will be randomly assigned (3:1) to receive either modified FOLFOX6 [mFOLFOX6] chemotherapy combined with Antigen Pulsed Dendritic Cells (Arm APDC + Chemotherapy), or chemotherapy alone (Arm Chemotherapy). Each patient recruited in the study will receive maximum 12 cycles of (14 days/cycle) mFOLFOX6 chemotherapy. Patients in Arm APDC + Chemotherapy will receive APDC vaccination in addition to chemotherapy in the cycle 1-3 and 7-9, and in cycle 4-6 and 10-12 receive only chemotherapy. APDC + Chemotherapy or Chemotherapy will be stopped in case of disease progression, intolerable toxicities, or patient withdrawal with the consent. After 12 cycles, patients in Arm APDC + Chemotherapy will receive 5-Fluorouracil treatment plus every 3 months APDC therapy and patients in Arm Chemotherapy will receive only 5-Fluorouracil treatment. PFS, ORR and OS will be assessed, and toxicity and immunologic effects will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the colorectum with metastatic lesions and received no previous therapy for metastatic lesions;
2. Be able to undergo surgical resection to obtain at least 1cm3 tumor tissues;
3. The patients are from 18-75 years old regardless of gender;
4. An estimated life expectancy of more than 6 months with ECOG≤2;
5. Adequate hepatic, renal, and bone marrow functions: neutrophilic granulocyte≥1.5×109/L, Hb(hemoglobin)≥90g/L, PLT(platelets)≥100×109/L, serum Cr(creatinine)≤1.5-time upper normal limit, serum TBIL(total bilirubin)≤1.5-time upper normal limit, both serum ALT and AST(alanine aminotransferase and aspartate aminotransferase)≤2.5-time upper normal limit, hepatic metastases CRC patients' serum ALT/AST≤5-time upper normal limit;
6. At least one measurable lesion after surgical resection (According to the standard of RECIST1.1 version: Response Evaluation Criteria in Solid Tumors 1.1 version);
7. Written informed consent.

Exclusion Criteria:

1. Severe (ie, active) heart disease, such as coronary heart disease symptoms, the New York Heart Association (NYHA) II-class or more serious congestive heart failure or severe arrhythmia requiring medication intervention, or history of myocardial infarction within the last 12 months; severe pulmonary dysfunction; peripheral neuropathy; unstable hypertension;
2. Metastases lesions> 50% of liver volume;
3. Autoimmune diseases, organ transplantation requiring immunosuppressive therapy and patients requiring long-term systemic corticosteroid therapy;
4. History of other malignant diseases (except cured basal cell carcinoma and cervical carcinoma in situ) in the last 5 years;
5. Pregnant or lactating women (women at childbearing age in the baseline pregnancy test positive or pregnancy test not examined. Menopausal women have menopause at least 12 months);
6. Acute or chronic infectious diseases in active phase; severe uncontrolled infection, or other serious uncontrolled concomitant diseases;
7. Definite history of allergy or allergic constitutions;
8. Chemotherapy, radiotherapy or immunotherapy within four weeks;
9. Administration of other investigational drugs or procedures within four weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival, PFS | Up to approximately six years
  Time from the randomization date to the start of disease progression (progression assessed by investigator using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1 guidelines) for metastatic colorectal cancer subjects.

SECONDARY OUTCOMES:
Objective Response | Up to approximately six years
  From randomisation to occurrence of objective response( complete regression (CR) and partial regression (PR) need to be confirmed 28 days after the occurrence)
Overall Survival, OS | Up to approximately six years
  From randomisation to the time of death of any cause.
Clinical benefit Rate | Up to approximately six years
  From randomisation to confirmation of objective response
Quality of Life | Up to approximately six months
  From randomisation to the end of all treatments (according to the EORTC QLQ-C30: European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire-C30)
Adverse Events | Up to approximately six years
  From randomisation to the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Xuetao Cao, M.D.,Ph.D., Study Chair — Second Military Medical University; Tao Wan, Ph.D., Study Director — Second Military Medical University; Yuankai Shi, M.D.,Ph.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences